CLINICAL TRIAL: NCT01779674
Title: Atrial Fibrillation/Sinus Rhythm Before and After Cardioversion
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-079
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study´s aim is to collect scientific data about patients with atrial inflammation by two principles of sensors measuring congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

* patients with atrial fibrillation and planned cardioversion
* male and female patients aged at least 18 years
* patients being able to understand and to follow the study staff´s instructions
* signed informed consent

Exclusion Criteria:

* persons being hosted in an institution by administrative order or court injunction
* pregnancy or breast feeding
* persons not being able to consent
* persons with implanted electronic devices
* material incompatiblity
* acute or chronic inflammation of the external or middle ear canal
* abnormal anatomic ear canal (congenital or pathological)
* persons in a dependent relationship to the investigator or employment contract

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
scientific data | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital Aachen, Aachen, North Rhine Westfalia, Germany

REFERENCES:
- [Derived] Zink MD, Bruser C, Winnersbach P, Napp A, Leonhardt S, Marx N, Schauerte P, Mischke K. Heartbeat Cycle Length Detection by a Ballistocardiographic Sensor in Atrial Fibrillation and Sinus Rhythm. Biomed Res Int. 2015;2015:840356. doi: 10.1155/2015/840356. Epub 2015 Jul 1. PMID 26229965